CLINICAL TRIAL: NCT05918926
Title: Salaso Moving More: The Impact of Digitally Delivered Precision Exercise in Helping People to Move More
Brief Title: Digitally Delivered Exercise in Helping People to Move More
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangor University (Other)
Collaborators: Betsi Cadwaladr University Health Board (Other Government); Salaso Health Solutions Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRAS300828
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2022-07

CONDITIONS: Obesity
Keywords: Physical activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Remote 12-week exercise intervention
  Interventions: Behavioral: Exercise
- Control/Routine Care (No Intervention): No exercise intervention, continue with routine care

INTERVENTIONS:
Behavioral: Exercise — Individualised remote exercise intervention
  Arms: Exercise

SUMMARY:
The main objective of this study is to examine the influence of the digital exercise prescription platform in increasing habitual physical activity in people on a weight management programme.

DETAILED DESCRIPTION:
Participants will be provided with individualised exercise training from exercise specialists. Participants will be recruited from the BCUHB NHS KindEating programme for people who have obesity (BMI of >30 kg/m2). Participants will be recruited remotely, via their KindEating dietitian. The assessments and exercise programme will be conducted remotely in the participants' own home.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled into the KindEating programme with BCUHB
* ≥ 18 years of age
* Able to provide written informed consent

Exclusion Criteria:

* Any uncontrolled medical condition that is exacerbated by exercise
* Unstable angina, unstable or acute heart failure, new or uncontrolled arrhythmias, resting or uncontrolled tachycardia, uncontrolled hypertension >180/100 (in either), symptomatic hypotension, febrile illness, acute uncontrolled psychiatric illness, other rapidly progressing terminal illness, uncontrolled diabetes >16.7mmol, patient's currently undergoing anti-biotic treatment for cellulitis, acute infections active foot ulceration
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Habitual physical activity | Change between baseline and 3 months (post intervention)
  Global Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sophie E Harrison, PhD, Principal Investigator — Bangor University
Locations (1):
- Betsi Cadwaladr University Health Board, Bangor, North Wales, United Kingdom